CLINICAL TRIAL: NCT00245700
Title: Study of Adherence of Stalevo, Entacapone and Levodopa
Brief Title: Adherence of Stalevo, Entacapone and Levodopa
Status: Completed | Type: Observational
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Responsible Party: Dr D Grosset, Southern General Hospital
Other Study IDs: R050017; Grant from Orion Pharma
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
To test if combining two antiparkinson drugs into a single tablet improves accuracy of medicine intake by the patient.

To test if patients with Parkinson's disease who take medicines at regular time intervals have smoother symptom control.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease aged between 18 and 85 years fulfilling UK Brain Bank criteria.
* Current levodopa therapy prescribed on a regular basis three or more times per day but requiring entacapone because of 'wearing off'
* Able to manipulate electronic monitoring bottles and complete questionnaires

Exclusion Criteria:

* Current use of compliance aid such that study participation would be detrimental to patient's adherence
* Pregnancy or breast feeding
* Excess alcohol (over 21 units per week for women and 28 units for men)
* Mini mental state examination of less than 26.
* Severe depression (Geriatric depression score over 20)

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2005-04; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald G Grosset, MBChB, MD, Principal Investigator
Locations (1):
- Southern General Hospital, Glasgow, Scotland, United Kingdom